CLINICAL TRIAL: NCT05393635
Title: A Phase 1, Open-Label, Multicenter Study Evaluating the Safety, Feasibility, and Preliminary Efficacy of ITIL-168 With Pembrolizumab in Subjects With Advanced Solid Tumors
Brief Title: ITIL-168 in Advanced Solid Tumors
Acronym: DELTA-2
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: business decision
Sponsor: Instil Bio (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITIL-168-102
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Cervical Cancer; Head and Neck Squamous Cell Carcinoma; Non-small Cell Lung Cancer
Keywords: ITIl-168; Cell Therapy; Cervical cancer; Head and neck squamous-cell carcinoma (HNSCC); Non-small cell lung cancer (NSCLC); Autologous Adoptive Cell Therapy; Cellular Immunotherapy; Immuno-oncology; Tumor Infiltrating Lymphocytes; TIL; T-cell therapy; IL-2; pembrolizumab; Checkpoint inhibitor (CPI); PD-1 pathway inhibitors
MeSH Terms: conditions — Uterine Cervical Neoplasms; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Participants with cervical cancer whose disease has progressed during or after treatment with platinum-based chemotherapy. Participants with combined positive score ≥ 1 should also have disease that has progressed during or after treatment with CPI.
  Interventions: Biological: ITIL-168
- Cohort 2 (Experimental): Participants with head and neck squamous-cell carcinoma (HNSCC) whose disease has progressed during or after platinum-based chemotherapy and previous CPI.
  Interventions: Biological: ITIL-168
- Cohort 3 (Experimental): Participants with non-small cell lung cancer (NSCLC) whose disease has progressed during or after platinum-based chemotherapy and a CPI. Participants with targetable mutations (e.g. EGFR/ALK) are required to have disease which has progressed on targeted therapy and platinum-based chemotherapy.
  Interventions: Biological: ITIL-168

INTERVENTIONS:
Biological: ITIL-168 — ITIL-168 is a cell therapy product derived from a participant's own TILs. A portion of tumor is resected to make a personalized ITIL-168 product. If appropriate, participants may receive bridging therapy after recovering from the tumor resection during ITIL-168 manufacturing. Once ITIL-168 has been made, the participant is treated with up to 5 days of lymphodepleting chemotherapy including cyclophosphamide and fludarabine, followed by a single infusion of ITIL-168, and up to 8 doses of IL-2.
  Drug: Pembrolizumab Participants will receive 1 dose of pembrolizumab following tumor resection prior to receiving ITIL-168, and additional doses for up to a year after ITIL-168 infusion.

SUMMARY:
DELTA-2 is a phase 1 clinical trial to evaluate the safety, feasibility, and preliminary efficacy of ITIL-168 with pembrolizumab in participants with advanced cancer whose disease has progressed after standard therapy. ITIL-168 is a cell therapy derived from a patient's own tumor-infiltrating immune cells (lymphocytes; TILs).

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically documented advanced (metastatic and/or unresectable) cervical cancer, HNSCC, or NSCLC.
* Cohort 1: Participants with cervical cancer whose disease progressed during or after at least 1 prior line of chemotherapy.
* Cohort 2: Participants with HNSCC whose disease progressed during or after chemotherapy that must have included a platinum agent and previous CPI.
* Cohort 3: Participants with NSCLC whose disease progressed during or after 1 prior line of platinum-based chemotherapy and a CPI. Participants with targetable mutations (e.g. EGFR/ALK) are required to have progressed on targeted therapy and platinum-based chemotherapy
* Medically suitable for surgical resection of tumor tissue
* Following tumor resection for TIL harvest, will have, at minimum, 1 remaining measurable lesion as identified by CT or MRI per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Adequate bone marrow and organ function

Key Exclusion Criteria:

* History of another primary malignancy within the previous 3 years
* Neuroendocrine carcinoma, nasopharyngeal carcinoma, squamous cell carcinoma of the lip, or histopathology with neuroendocrine differentiation
* Previously received an allogeneic stem cell transplant or organ allograft
* Previously received TIL or engineered cell therapy (eg, CAR T-cell)
* Significant cardiac disease
* Stroke or transient ischemic attack within 12 months of enrollment
* History of significant central nervous system (CNS) disorder
* Symptomatic and/or untreated CNS metastases
* History of significant autoimmune disease within 2 years prior to enrollment
* Known history of severe, immediate hypersensitivity reaction attributed to cyclophosphamide, fludarabine, IL-2, of CPI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08 (Estimated); Primary Completion 2022-12-08 (Actual); Study Completion 2022-12-08 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of ITIL-168 treatment-emergent adverse events (AEs), serious AEs, and AEs of special interest | Up to 24 months

SECONDARY OUTCOMES:
Objective response rate | Up to 60 months
  Objective response rate (ORR), defined as the incidence of a complete response (CR) or a partial response (PR) per a modified Response Evaluation Criteria in Solid Tumors (RECIST v1.1) criteria, as assessed by investigator review.
Duration of response | Up to 60 months
  For participants who experience an objective response, duration of response (DOR) is defined as the time from their first objective response to disease progression or death.
Progression-free Survival | Up to 60 months
  Progression-free survival (PFS) is defined as the time from the ITIL-168 infusion date to the date of disease progression or death from any cause.
Overall Survival | Up to 60 months
  Overall survival (OS) is defined as the time from the ITIL-168 infusion date to the date of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Instil Study Director, Study Director — Instil Bio, Inc.

IPD SHARING:
Plan to Share IPD: No